CLINICAL TRIAL: NCT04315610
Title: Personalized Mobile App for Parents of Infants With Cardiac Disease
Acronym: HOBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Association for Children with Congenital Heart Disease (FFHB) (Unknown)
Responsible Party: Principal Investigator, Henrik Holmstrøm, Professor, Oslo University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 19/23041
Record Dates: First submitted 2019-10-16; First posted 2020-03-19 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Disease in Children; Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to mobile application (Experimental): This application will help parents to recognize symptoms of reduced health status in their infant, provide decision-making support, increase their communication skills with health professionals, and provide easier access to quality assured information. At first login, the diagnosis, treatment, and contacts in the health service are registered to provide parents with personalized information that is adapted to their infant's needs. Under the guidance of healthcare personnel at the Neonatal Intensive Care Department (NICD) at Oslo University Hospital (OUH), parents are trained to assess their infant's condition, regarding circulation, breathing, eating habits, well-being, and more. In addition, before discharge, a baseline assessment of the infant's condition is stored in the application.
  Interventions: Other: Access to mobile phone application
- Treatment as usual (Active Comparator): This group receives traditional oral and written information about their child's heart defect and further follow-up.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Access to mobile phone application — Under the guidance of healthcare personnel at the Neonatal Intensive Care Department (NICD) at Oslo University Hospital (OUH), parents are trained to assess their infant's condition, regarding circulation, breathing, eating habits, well-being, and more. In addition, before discharge, a baseline assessment of the infant's condition is stored in the application. After discharge, assessments using the application are performed if necessary.
  Arms: Access to mobile application
Other: Treatment as usual — Active comparator group, based on traditional information and follow-up.
  Arms: Treatment as usual

SUMMARY:
This project implements an eHealth intervention targeted at vulnerable infants with cardiac disease and specifically study how this intervention impact their parents coping, stress levels and personal wellbeing. The intervention will be evaluated through a pragmatic controlled trial.

The aim of this project is therefore to measure if the features of this mobile application are useful for parents' assessment of deterioration, decision-making and communication with health care providers.

DETAILED DESCRIPTION:
This project is a service innovation project where the overall aim is to stimulate service innovation that ensures patient safety to vulnerable infants with severe cardiac disease. We plan to implement and evaluate an eHealth intervention, called HOBS (the Heart OBServation-app), that systemizes and personalizes information and teaching from nurses and other health personnel in order to support parents as caregivers after discharge from hospital. The service innovation will be studied in two consecutive studies; 1) a feasibility study to examine health personnel and parents in-depth perception of relevance, benefit and user friendliness of the application and its features, and 2) a controlled trial to measure the applications impact on parents stress, anxiety, coping and health literacy after discharge, including reasons and outcomes of contact with health services. In addition, we evaluate if nurses' quality of discharge teaching is affected by the application.

In Norway, 500-600 children are born with congenital heart defects (CHD) every year. About 25% of these children present severe problems and symptoms in need of early treatment (1), and 15 % of them die during the first year of life (2). Parents of infants with cardiac disease assume significant, comprehensive caregiving responsibilities, and have shown higher levels of anxiety, depression, and stress. Many parents find it difficult to recognize the symptoms if their child's health and wellbeing deteriorates(3).

New, mobile technology applications and services come with novel opportunities to support these parents with personalized, contextual information at the point of need. For example, interactive functions and presentation of selected information can enable personalized decision-making and communication support. This can improve relevance and quality of discharge teaching from nurses at Neonatal Intensive Care Department (NICD) at Oslo University Hospital (OUH), but more importantly also support local services where CHD seldom occur and knowledge may be sparse. To date, the value added, appropriateness and importance of such opportunities for mental stress and health competence among parents of children with CHD has not been systematically reported. Moreover, if our study goals are achieved, the intervention can empower parents to recognize the early signs before deterioration in their infant manifests, prevent acute episodes at home after discharge, and improve rehabilitation. For the parents this service innovation may reduce psychological strain during a challenging period of life.

Method and data collection A controlled trial with consecutive groups has been chosen to avoid contamination of health personnel's way of guiding and parents interaction at common rooms at the NICD. Even though the access to or use of the application are controlled by the project using a login code we accept that guidance will be affected and more systematic during the implementation of the application and this may affect the results. Hence, a two months break between the last family receiving app in the quality study at OUH and inclusion of the control group is planned. Inclusion of the control group will then be conducted before inclusion of the app group. The control group receives written information in a binder while the intervention group will receive the information through links in the mobile application. A guideline including a checklist of topics to support parents before discharge is similar to both groups.

The intervention HOBS-app is developed by a project group at OUH together with parents and local health personnel for parents with infants with cardiac disease. It is presented in detail at the web-page www.hobs.no. Congenital heart disease is a complicated and individual diagnosis with varied consequences (15). Therefore, at first login, the diagnosis and treatments are registered. Then an algorithm in the application provides parents with a personalized set of observations and a list of adapted information to their infant's needs. Under the guidance of nurses at the NICD at OUH, parents are trained using the app to assess their infant's condition, regarding circulation, breathing, eating habits, well-being, wound healing and more. These observations are stored in the application. In this way parents become better aware of their infant's condition and may help parents to detect signs of deterioration at home. Contact information to local health services is stored before discharge. After discharge, assessments using the application are performed before consultations to health services or if parents are uncertain about deterioration in their infant. After assessments the applications' function for communication support can guide parents in describing a possible deterioration and communication with health personnel may be facilitated.

To reach health professionals with information about HOBS a website will be established with guidance and tips on using the app. An e-learning course is developed and will be distributed nationally through similar educative portals. A link to the website and the e-learning courses are added to the discharge summary that follows the infant to a local hospital.

The purpose of the controlled trial is to answer research question 3: In what ways do the application's content and functionality influence the parents' coping with stress, anxiety, distress of caring for a sick child and health literacy and contact with health services?

ELIGIBILITY:
Inclusion Criteria:

Infants below 3 months age diagnosed with severe heart disease at NICD at OUH

Exclusion Criteria:

a) Gestational age below 34 weeks b) Isolated arrhythmic disorders c) Language barriers d) Need of advanced home care with professional assistance

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Pediatric Inventory for Parents (PIP) | Baseline, 1 and 4 months
  The PIP measures parental stress related to children with chronic disease and is the primary endpoint regarding psychological adaption. It contains 42 items that are answered on a 5-point Likert scale within four domains: 1) communication, 2) emotional distance, 3) medical care and 4) role function. All items are answered twice, one for frequency and one for difficulty. Higher score reflects more disease-related stress. The instrument has shown good reliability and content validity. The instrument can provide answers about the causes and degree of stress and anxiety. The instrument has been translated into Norwegian using acknowledged methods.

SECONDARY OUTCOMES:
Health literacy Questionnaire (HLQ) | 4 months
  The HLQ is a multidimensional instrument that measures health competence and has good validity and reliability. It consists of nine areas within health competence, and a selection can be made based on the intervention's objective (42). The following four scales will be used in this study (number from original questionnaire in parentheses): (6) ability to interact with health professionals, (7) orientation in health care, (8) ability to find good health information, and (9) understanding health information in order to know what action to take. In total, 20 items will be answered. The instrument is translated into Norwegian and has been subject to psychometric assessment in an adult population. Scores range between 1 to 4 (for first 5 scales) and 1 to 5 (for scales 6 to 9), and higher value indicates better literacy.
Post Discharge Coping Difficulty Scale (PDCDS) | 1 month
  PDCDS measures parental coping after discharge and is the primary outcome after 1 month. It has good reliability and validity. The instrument is translated in to Norwegian and has acceptable reliability (0.71) (18) . The scale uses an 11 point format with anchor words ("not at all" to "totally") at the 0 and 10 poles of the scale, where higher value indicates more difficulties. Five of the questions have an additional open ended question that elaborates what kind of difficulties parents' experience.
Edinburgh postnatal depression scale (EPDS) | Baseline, 1 and 4 months
  The EPDS is a self-rating scale developed to screen for postnatal depression. It consists of 10 items. Each statement has four possible responses, which are scored from 0 to 3, depending on the severity of the response. Higher scores indicate more severe depressive symptoms with a maximum total score of 30. It has been translated into Norwegian with good reliability: Cronbach's alpha of 0.89. Depression is a common challenge among parents of infants with CHD, and it may affect other dependent outcomes like PIP and perception of coping and knowledge in the study.
Quality of discharge teaching scale (QDTS) | At discharge from local hospital (up to 5 days)
  The QDTS consists of 18 items using a similar format as the RHDS, with two subscales and questions about the information given by nurses. It has good reliability and validity (34). The instrument is translated into Norwegian and has demonstrated good reliability, with Cronbach's alpha of 0.89. The content subscale consists of six paired items where parents assess needed and received information regarding preparation for discharge. The second subscale consists of 12 items and reflects nurses' skills as educators. This instrument detected significantly increased content of information in parents of infants with CHD receiving written information compared to standard oral information in 2013.
Readiness for hospital discharge (RHDS) | At discharge from local hospital (up to 5 days)
  The RHDS is based on transition theory. It measures parents' perception of readiness for hospital discharge and is the primary outcome at discharge. It consists of 23 items and has good validity and reliability. It has been translated into Norwegian. It contains four subscales regarding discharge preparedness: 1) parent and child personal status, 2) knowledge, 3) coping ability and 4) expected support. The scale uses an 11-point format with anchor words ("not at all" and "totally") at the 0 and 10 poles of the scale. Our hypothesis is that higher availability of information and more systematic observations of the infant's appearance will increase perception of readiness and knowledge compared to standard care.
User log and additional questions | From inclusion until 4 months
  To observe parents' use of HOBS, log data about use will be extracted. This includes settings at discharge, time and frequency of assessments of the infant and use of information links. The log data can illuminate user patterns, which features are most used and how use of HOBS changes over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hjorth-Johansen E, Borosund E, Martinsen Osten I, Holmstrom H, Moen A. Acceptability and Initial Adoption of the Heart Observation App for Infants With Congenital Heart Disease: Qualitative Study. JMIR Form Res. 2023 Apr 5;7:e45920. doi: 10.2196/45920. PMID 37018028
- [Background] Hjorth-Johansen E, Borosund E, Moen A, Harmens A, Martinsen I, Wik G, Fredriksen BE, Eger SHW, Holmstrom H. Heart OBServation app: development of a decision support tool for parents of infants with severe cardiac disease. Cardiol Young. 2023 Aug;33(8):1350-1358. doi: 10.1017/S1047951122002438. Epub 2022 Aug 8. PMID 35938297
- [Result] Hjorth-Johansen E, Borosund E, Moen A, Osten IM, Wik G, Solevag AL, Eger SHW, Holmstrom H. An individualised mobile app was beneficial for the mothers of infants with severe congenital heart defects. Acta Paediatr. 2025 Jun;114(6):1238-1248. doi: 10.1111/apa.17556. Epub 2024 Dec 21. PMID 39707745